CLINICAL TRIAL: NCT06381778
Title: Taiwan Registry of Hypertrophic Cardiomyopathy (THIC) Research Synopsis
Status: Recruiting | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yen-Wen Wu, Director, Cardiovascular Medical Center, Far Eastern Memorial Hospital, Far Eastern Memorial Hospital
Other Study IDs: 112006-E
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypertrophic cardiomyopathy (HCM) is hallmarked by the presence of left ventricular hypertrophy (LVH) and may present various symptoms including arrhythmia and heart failure. Mutations in the genes related to sarcomeric proteins and metabolic disorders are known causes of HCM. However, it remains required to further explore the prevalence of HCM in the context of Taiwanese' genetic background. Additionally, certain rare diseases that affect the heart, including Fabry disease, cardiac amyloidosis, may present LVH, which makes precise diagnosis among HCM and these diseases more challenging. In this TSOC multi-center registry, we aim to systematically evaluate the clinical, genetic, biochemical features,prevalence, and possible natural course of HCM and relevant rare diseases such as Fabry disease in Taiwan. In the meanwhile, we may also generate the specific "red-flag" signs of Fabry disease in Taiwan.

DETAILED DESCRIPTION:
Hypertrophic cardiomyopathy (HCM) is hallmarked by the presence of left ventricular hypertrophy (LVH) . Studies across geographic areas report a prevalence of unexplained LVH at 0.02-0.23% in adults, and a trend of age-related prevalence, with lower rates in patients under the age of 25 years . HCM may present in a wide variety of patterns. Its natural history includes the development of progressive, life-limiting symptoms due to left ventricular outflow tract (LVOT) obstruction or diastolic dysfunction, atrial arrhythmias, heart failure (HF) associated with systolic dysfunction and risk of ventricular arrhythmias. HCM is frequently transmitted in an autosomal dominant manner. Known etiologies include mutations in the genes related to sarcomeric proteins, metabolic disorders, neuromuscular diseases, and inflammation. The good prognosis depends on early diagnosis and correct treatment strategy.

Fabry disease (FD) is an X-linked rare disease caused by mutations in the GLA gene, which encodes alpha-galactosidase A (alpha-GAL A). Defects in alpha-GAL A leads to accumulation of Gb3 in cells, which in turn impairs the function tissues and organs. Different GLA variants may be related to various symptoms in different organs, and these variants can be categorized into two types: classic and late-onset. In classic type of patients, the disease manifestations usually occur in childhood with common symptoms such as extremity pain, nausea, fever of unknown origin and hypohidrosis. In addition, classic FD patient may present renal and cardiac deteriorations as well as cerebrovascular manifestations. These manifestations may further develop into life-threatening complications at middle or late age if untreated [4]. On the other hand, disease onset in late-onset type of FD patients is typically in adulthood, and the clinical manifestations may be limited to fewer organs compared to what was found in the classic type. For example, cardiac variants IVS4+919G>A and p.N215S tend to affect the heart. Because cardiac abnormalities in FD such as LVH is like what is observed in several heart conditions such as HCM and cardiac amyloidosis, differential diagnosis between FD and other heart conditions is a topic of great research and clinical interest.

Although LVH is a common feature between FD and HCM, the prevalence of FD in HCM patients is usually limited to 1-2%. Hence, several recent reports strive to describe the development of criteria to increase the accuracy of diagnosis of FD in HCM/LVH populations. Seo et al. prospectively assessed the cardiac screening criteria to increase the chance of identification of FD in HCM patients via integration of data on short PR interval, arrhythmia, and symptoms of autonomic function. In addition, Fan et al. focused on patients with IVST or PWT ≥ 13 mm on echocardiography, and excluded patients with known sarcomeric gene mutations, amyloidosis, athletic heart, non-compaction cardiomyopathy, and non-FD metabolic or syndromic conditions associated with LVH. However, these reports are limited to single or very few centers. Moreover, it needs to be cautious to interpret these study results due to various distribution of FD mutations in different countries or geographic areas.

On the other hand, amyloid deposition in the heart is called cardiac amyloidosis (CA); 95% is immunoglobulin light chain amyloidosis (AL) and transthyretin amyloidosis (ATTR). Hereditary (ATTRm) or wild-type (ATTRwt) depends on whether the ATTRm gene is mutated or not. The most common mutation in Taiwan is A97S, 80% have LVH. And bone-avid tracers such as 99mTc-PYP/DPD/HMDP could detect CA, which may be related to the microcalcification. Recent advances in therapeutic strategies shown to be most beneficial in the early stages of the disease have determined a paradigm shift in the screening, diagnostic algorithm, and risk classification of patients with ATTR-CM.

Patients with HCM have genotypic and phenotypic variability. There are a number of treatment modalities for these patients, including pharmacotherapy to control symptoms, implantable cardiac defibrillators to manage malignant arrhythmias, and surgical myectomy and septal ablation to decrease the left ventricular outflow obstruction. Accurate diagnosis is vital for the perioperative management of these patients. Of note, other LVH conditions such as FD, CA also have specific genetic background in Taiwan. In this program, Taiwan Socieyt of Cardiology aims to establish a multi-center registry that includes FD and selected heart conditions featured by unexplained LVH. This registry will allow understanding of the clinical features and disease patterns of patients with unexplained LVH in Taiwan. With systematic documentation of features of FD and non-FD patients across Taiwan, this registry might serve as an asset for future research such as development of scoring algorithm to identify FD more precisely, and generate the specific "reg-flag" signs in FD, in comparison with HCM or CA in Taiwan. Moreover, with documentation of clinical and biochemical parameters and clinical follow-up, this registry will allow future research to understand the natural history of FD or HCM, and long-term treatment outcomes of these diseases in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of left ventricular hypertrophy (LVH) on echo/CMRI:
2. maximal interventricular septal (IVST) and/or posterior wall thickness (PWT) ≥13 mm,
3. apical wall thickness ≥15 mm or a ratio of apical to basal LV wall thickness of ≥ 1.3 at end-diastole, OR
4. maximal LV wall thickness ≥ 15mm of ANY OTHER PART
5. Male and female adult age ≥ 20 year-old
6. Patients willing to comply with and sign the informed consent

Exclusion Criteria:

1. Patients refuse or unable to give informed consent
2. Patients unlikely to comply with the protocol or unable to understand the nature and possible consequences of the program
3. Co-arctation of the aorta, severe aortic stenosis, or severe LV pressure overload
4. Athletic heart
5. Non-compaction cardiomyopathy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Presence of left ventricular hypertrophy
Sampling Method: Probability Sample
Enrollment: 2600 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Death | 1 year
  Death

SECONDARY OUTCOMES:
CV death | 1 year
  CV death

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No